CLINICAL TRIAL: NCT06192108
Title: A Phase 3, Randomized, Open-Label Study to Investigate the Efficacy and Safety of Once Daily Oral Orforglipron Compared With Dapagliflozin in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Metformin (ACHIEVE-2)
Brief Title: A Study of Orforglipron (LY3502970) Compared With Dapagliflozin in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Metformin
Acronym: ACHIEVE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18566; J2A-MC-GZGV (Other: Eli Lilly and Company); 2023-507206-13-00 (Other: EU Trial Number); U1111-1296-1507 (Other: UTN Number)
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — orforglipron; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Orforglipron Dose 1 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 2 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Orforglipron Dose 3 (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Dapagliflozin (Active Comparator): Participants will receive dapagliflozin orally.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
  Arms: Orforglipron Dose 1; Orforglipron Dose 2; Orforglipron Dose 3
Drug: Dapagliflozin — Administered orally
  Arms: Dapagliflozin

SUMMARY:
The main purpose of this study is to assess the safety and efficacy of orforglipron compared with dapagliflozin in improving blood sugar control in participants with type 2 diabetes (T2D) with inadequate glycemic control using metformin. The study will last approximately 46 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of T2D based on the World Health Organization classification or other locally applicable diagnostic standards.
* Have HbA1c ≥7.0% (53 mmol/mol) to ≤10.5% (91 mmol/mol) at screening.
* Have been on stable diabetes treatment with metformin ≥1500 milligram per day (mg/day) during the 90 days prior to screening and maintained through randomization.
* Are of stable body weight (±5%) for at least 90 days prior to screening and agree to not initiate an intensive diet or exercise program during the study with the intent of reducing body weight, other than the lifestyle and/or dietary measures for diabetes treatment.
* Have a body mass index (BMI) ≥23.0 kilogram/square meter (kg/m²) at screening.

Exclusion Criteria:

* Have Type 1 Diabetes (T1D)
* Are currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema
* Have an estimated glomerular filtration rate (eGFR) <45 milliliter per minute (mL/min)/1.73 square meter (m2)
* Have acute or chronic hepatitis
* Have had chronic or acute pancreatitis any time.
* Have been treated with any antihyperglycemic medication (other than metformin) within the 90 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 962 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c: (HbA1c) | Baseline, Week 40

SECONDARY OUTCOMES:
Change from Baseline in HbA1c | Baseline, Week 40
Percentage of Participants Who Achieved HbA1c <7.0% (53 millimole/mole(mmol/mol)) | Week 40
Percentage of Participants Who Achieved HbA1c ≤6.5% (48 mmol/mol) | Week 40
Percentage Change from Baseline in Body Weight | Baseline, Week 40
Change from Baseline in Body Weight | Baseline, Week 40
Percentage Change from Baseline in Non-High-Density Lipoprotein (non-HDL)-Cholesterol | Baseline, Week 40
Percentage Change from Baseline in Triglycerides | Baseline, Week 40
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 40
Change from Baseline in Fasting Serum Glucose | Baseline, Week 40
Percentage of Participants Who Achieved Weight Loss of ≥5% from Baseline | Baseline to Week 40
Percentage of Participants Who Achieved Weight Loss of ≥10% from baseline | Baseline to Week 40
Percentage of Participants Who Achieved Weight Loss of ≥15% from baseline | Baseline to Week 40
Change from Baseline in Diastolic Blood Pressure (DBP) | Baseline, Week 40
Percentage Change from Baseline in Total Cholesterol | Baseline, Week 40
Change from Baseline in Short Form 36 Version 2 (SF-36-v2) Acute Form Domain Summary Scores | Baseline, Week 40
Change from Baseline in Diabetes Treatment Satisfaction Questionnaire-Change (DTSQc) Scores | Baseline, Week 40

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (74):
- United States (19):
  - Alliance Research Institute - Canoga Park, Canoga Park, California
  - Ark Clinical Research, Long Beach, California
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California
  - Wolverine Clinical Trials, Santa Ana, California
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Institute of Endocrinology Diabetes, Health & Hormone, Stockbridge, Georgia
  - Elite Clinical Trials, Rexburg, Idaho
  - Accellacare - DuPage, Lombard, Illinois
  - Tandem Clinical Research, Marrero, Louisiana
  - St. Vincent Healthcare, Billings, Montana
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Accellacare - Winston-Salem, Winston-Salem, North Carolina
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Essential Medical Research, Tulsa, Oklahoma
  - Accellacare - Mt Pleasant, Mt. Pleasant, South Carolina
  - Accellacare, US Inc., d/b/a Accellacare of Knoxville, Jefferson City, Tennessee
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Juno Research, Houston, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
- China (12):
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Germany (11):
  - CRS Clinical Research Services Mannheim, Mannheim, Baden-Wurttemberg
  - Diabetologische Schwerpunktpraxis Dr. Staudenmeyer & Dr. Schiwietz, Lingen, Lower Saxony
  - Diabetes- und Stoffwechselpraxis Bochum, Bochum, North Rhine-Westphalia
  - Zentrum fur klinische Forschung - Köln, Cologne, North Rhine-Westphalia
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Medizentrum Essen Borbeck, Essen, North Rhine-Westphalia
  - Institut für Diabetesforschung GmbH Münster, Münster, North Rhine-Westphalia
  - Praxis Dr. Veronika Wenzl-Bauer, Rehlingen, Saarland
  - Zentrum für klinische Studien, Saint Ingbert, Saarland
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Diabetes Zentrum Wilhelmsburg, Hamburg
- Mexico (13):
  - Grupo Ollin Care, Pachuca, Hidalgo
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, Guadalajara, Jalisco
  - Cryptex Investigación Clínica S.A. de C.V., Cuauhtémoc, Ciudad de México, Mexico City
  - ProcliniQ Investigación Clínica SA de CV, Mexico City, Mexico City
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca, Morelos
  - Cardiolink Clin Trials, Monterrey, Nuevo León
  - Clínica García Flores SC, Monterrey, Nuevo León
  - Servicios Integrales Nova de Monterrey S.A. de C.V., San Nicolás de los Garza, Nuevo León
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán, Sinaloa
  - Consultorio de Medicina Especilizada del Sector Privado, Xalapa, Veracruz
  - Hospital Angeles Xalapa, Xalapa, Veracruz
  - Fundación Cardiovascular de Aguascalientes A.C., Aguascalientes
  - Lahoja. Asociacion Para La Investigacion Y La Farmacovigilancia, Durango
- Poland (11):
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow, Lesser Poland Voivodeship
  - Centrum Badań Klinicznych Piotr Napora lekarze sp.p., Wroclaw, Lower Silesian Voivodeship
  - Clinical Best Solutions, Lublin, Lublin Voivodeship
  - CenterMed Lublin NZOZ, Lublin, Lublin Voivodeship
  - Ekamed, Lublin, Lublin Voivodeship
  - Centrum Medyczne "Diabetika", Radom, Masovian Voivodeship
  - Zdrowie Osteo-Medic, Bialystok, Podlaskie Voivodeship
  - Specderm Poznanska, Bialystok, Podlaskie Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 1 SUM, Zabrze, Silesian Voivodeship
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz, Łódź Voivodeship
- Taiwan (8):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Fu Jen Catholic University Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Orforglipron (LY3502970) Compared With Dapagliflozin in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Metformin (ACHIEVE-2) — https://trials.lilly.com/en-US/trial/448175